CLINICAL TRIAL: NCT00045695
Title: A Phase II Study Of PS-341 (NSC 681239) In Patients With Untreated Or Relapsed Waldenstrom's Macroglobulinemia
Brief Title: Bortezomib in Treating Patients With Waldenstrom's Macroglobulinemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NCIC Clinical Trials Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); Eastern Cooperative Oncology Group (Network)
Responsible Party: Sponsor
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I152; CAN-NCIC-IND152; ECOG-JI152; NCI-NCIC-152; CDR0000257042 (Other: PDQ)
Record Dates: First submitted 2002-09-06; First posted 2003-01-27 (Estimated); Last update posted 2013-05-17 (Estimated); Status verified 2011-09

CONDITIONS: Lymphoma
Keywords: Waldenstrom macroglobulinemia
MeSH Terms: conditions — Lymphoma; Waldenstrom Macroglobulinemia | interventions — Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: bortezomib — PS-341 bolus intravenous injection twice weekly* for 2 out of every 3 weeks

SUMMARY:
RATIONALE: Bortezomib may stop the growth of cancer by blocking the enzymes necessary for tumor cell growth.

PURPOSE: Phase II trial to study the effectiveness of bortezomib in treating patients who have untreated or relapsed Waldenstrom's macroglobulinemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the efficacy of bortezomib, in terms of response rate, in patients with previously untreated or relapsed Waldenstrom's macroglobulinemia.
* Determine the toxicity of this drug in these patients.
* Determine the time to progression, stable disease duration, and response duration in patients treated with this drug.

OUTLINE: This is a multicenter study.

Patients receive bortezomib IV over 3-5 seconds on days 1, 4, 8, and 11. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Patients are followed at 4 weeks. Patients with complete or partial response or stable disease are followed every 3 months thereafter.

PROJECTED ACCRUAL: A total of 15-25 patients will be accrued for this study within 1.5-2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of Waldenstrom's macroglobulinemia confirmed by immunofixation or immunoelectrophoresis

  * Newly diagnosed or untreated with IgM ≥ 20 g/L OR
  * Previously treated with IgM ≥ 5 g/L
* Non-refractory, defined as no disease progression during prior therapy or within 4 weeks of the last dose of most recent prior therapy (12 weeks for rituximab)
* Must have 1 or more of the following:

  * Symptomatic lymphadenopathy
  * Hepatomegaly and/or splenomegaly
  * Anemia (i.e., hemoglobin < 11.0 g/dL)
  * Hyperviscosity syndrome
* No other lymphoproliferative disease including transformed aggressive lymphoma

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* At least 12 weeks

Hematopoietic

* See Disease Characteristics
* Absolute granulocyte count ≥ 1,000/mm^3
* Platelet count ≥ 50,000/mm^3

Hepatic

* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* AST or ALT ≤ 2.5 times ULN

Renal

* Creatinine ≤ 1.5 times ULN

Other

* No uncontrolled bacterial, fungal, or viral infection
* No pre-existing sensory or motor neurotoxicity grade 2 or greater
* No other prior malignancy except adequately treated nonmelanoma skin cancer, curatively treated carcinoma in situ of the cervix, or other curatively treated solid tumor for which patient has been disease free for at least 5 years
* No other serious illness or medical condition that would preclude study participation
* No unreasonable geographical limitations
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy

* See Chemotherapy
* See Disease Characteristics
* At least 12 weeks since prior rituximab (for patients who have progressed)
* At least 24 weeks since prior rituximab (for patients who have not progressed)
* No prior high-dose chemotherapy and stem cell transplantation
* No prior radioactive monoclonal antibodies

Chemotherapy

* See Disease Characteristics
* See Biologic therapy
* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin)
* No more than 2 prior chemotherapy regimens

  * The same chemotherapy combination given for first-line and second-line therapy is considered 2 regimens
  * Single-agent rituximab not considered 1 prior regimen
* No concurrent cytotoxic chemotherapy

Endocrine therapy

* No concurrent corticosteroids

Radiotherapy

* At least 4 weeks since prior radiotherapy (except for low-dose, non- myelosuppressive radiotherapy) and recovered
* No prior radiotherapy to more than 25% of bone marrow

Surgery

* At least 4 weeks since prior major surgery

Other

* At least 4 weeks since prior plasmapheresis
* At least 4 weeks since prior investigational anticancer therapy
* No other concurrent investigational anticancer agents or therapies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2002-08; Primary Completion 2006-03 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Response rate | 4 years
  To assess the efficacy (response rate) of PS-341 given as a bolus intravenous injection twice weekly for two out of every 3 weeks in the treatment of a population of patients with previously untreated or relapsed Waldenström's Macroglobulinemia

SECONDARY OUTCOMES:
Toxicity | 4 years
  To assess the toxicity of PS-341 in patients with Waldenström's Macroglobulinemia as well as time to progression, stable disease duration and, if responses are observed, response duration.
Cytogenetics and genome profiling | 4 years
  To assess bone marrow and peripheral blood for cytogenetics and genome profiling by microarray in patients with Waldenstrom's macroglobulinemia.

CONTACTS AND LOCATIONS:
Overall Officials: Christine I. Chen, MD, Study Chair — Princess Margaret Hospital, Canada
Locations (12):
- United States (2):
  - Hinsdale Hematology Oncology Associates, Hinsdale, Illinois
  - Abramson Cancer Center at the University of Pennsylvania, Philadelphia, Pennsylvania
- Canada (10):
  - Tom Baker Cancer Centre - Calgary, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Nova Scotia Cancer Centre at Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia
  - Margaret and Charles Juravinski Cancer Centre, Hamilton, Ontario
  - Cancer Care Ontario-London Regional Cancer Centre, London, Ontario
  - Toronto Sunnybrook Regional Cancer Centre, Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - Maisonneuve-Rosemont Hospital, Montreal, Quebec
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan

REFERENCES:
- [Result] Chen CI, Kouroukis CT, White D, Voralia M, Stadtmauer E, Stewart AK, Wright JJ, Powers J, Walsh W, Eisenhauer E; National Cancer Institute of Canada Clinical Trials Group. Bortezomib is active in patients with untreated or relapsed Waldenstrom's macroglobulinemia: a phase II study of the National Cancer Institute of Canada Clinical Trials Group. J Clin Oncol. 2007 Apr 20;25(12):1570-5. doi: 10.1200/JCO.2006.07.8659. Epub 2007 Mar 12. PMID 17353550
- [Result] Chen CI, White Darrell, Kouroukis TC, et al.: Antitumor activity of bortezomib (PS-341; Velcade) in a phase II study of patients with previously untreated or treated Waldenstrom's macroglobulinemia (WM). [Abstract] Blood 104 (11): A-3278, 2004.